CLINICAL TRIAL: NCT04647370
Title: Implications of Remote Ischemic Preconditioning on Liver Function in Adults Undergoing Cardiac Surgery: Randomized Controlled Trial
Brief Title: Remote Ischemic Preconditioning in Cardiac Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mostafa Samy Abbas, associate professor of anesthesia, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Ischemic Preconditioning
Record Dates: First submitted 2020-09-27; First posted 2020-11-30 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Ischemia Reperfusion Injury
MeSH Terms: conditions — Reperfusion Injury

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remote ischemic preconditioning (Active Comparator)
  Interventions: Procedure: remote ischemic preconditioning
- Sham remote ischemic preconditioning (Sham Comparator)
  Interventions: Procedure: Sham remote ischemic preconditioning

INTERVENTIONS:
Procedure: remote ischemic preconditioning — 3 cycles of 5-minutes inflation of a blood pressure cuff to 200mmHg (or at least to a pressure 50mm Hg higher than the systolic arterial pressure) to one upper arm, followed by5-minutes reperfusion with the cuff deflated
  Arms: Remote ischemic preconditioning
Procedure: Sham remote ischemic preconditioning — 3cycles of upper limb pseudo ischemia (low pressure, 5-minutes blood pressure cuff inflation to a pressure of 20 mm Hg and 5-minutes cuff deflation).
  Arms: Sham remote ischemic preconditioning

SUMMARY:
Aim of the work :

Evaluation of the role of Remote Ischemic Preconditioning (RIP) on liver function in patients undergoing on-pump cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Being candidate for on-pump cardiac surgery.
2. Willing to participate in the study
3. Ages eligible for the study: 18 to 70 years.
4. Gender eligible for the study : both

Exclusion Criteria:

1. Patient refusal.
2. Known cause of possible liver function disturbances that includes right heart failure, acute inflammation of gallbladder or any other complication of gallstone disease.
3. Active viral and non viral hepatitis.
4. Pregnant women.
5. History of peripheral nerve disease or peripheral vascular disease of the extremities

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
liver function test | 3 postoperative days
  Direct Bilirubin

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University hospital, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No